CLINICAL TRIAL: NCT06096103
Title: A Randomized, Double-blind, Parallel, Three-arms, Placebo-controlled, Safety and Efficacy Study of Botanical Extract Standardized for Iron + Vitamin C and Botanical Extract Standardized for Iron in Adult Human Subjects with Anemia or Iron-deficiency Anemia
Brief Title: A Clinical Study to Check the Safety and Effectiveness of Botanical Extract Standardized for Iron + Vitamin C and Botanical Extract Standardized for Iron in Adult Human Subjects with Anemia or Iron-deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Orgenetics, Inc. (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator- Medical Director, NovoBliss Research Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NB230024-OI
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2023-11

CONDITIONS: Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Parallel, Three-Arms, Placebo-Controlled
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) The study is double blind wherein neither the subjects nor the Investigator shall be aware of the test treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Take the test treatment once a day with food
  Interventions: Dietary Supplement: placebo
- Botanical Extract Standardised for Iron + Vitamin C (Experimental): The botanical extract standardised for iron and vitamin c is specially formulated for iron deficiency anaemia or anaemia. Vitamin C can promote the Iron absorption
  Interventions: Dietary Supplement: Botanical Extract Standardized for Iron + Vitamin C
- Botanical Extract Standardised for Iron (Experimental): The botanical extract standardised for iron is formulated for iron deficiency anaemia or anaemia
  Interventions: Dietary Supplement: Botanical Extract Standardised for Iron

INTERVENTIONS:
Dietary Supplement: placebo — Route: Oral Dosage: 500mg Dosage Form: Capsule Frequency: Once a Day Duration: 60 Days Mode of Usage: Take the capsule once a day with food
  Arms: Placebo
Dietary Supplement: Botanical Extract Standardized for Iron + Vitamin C — Route: Oral Dosage: 500mg Dosage Form: Capsule Frequency: Once a Day Duration: 60 Days Mode of Usage: Take the capsule once a day with food
  Arms: Botanical Extract Standardised for Iron + Vitamin C
Dietary Supplement: Botanical Extract Standardised for Iron — Route: Oral Dosage: 500mg Dosage Form: Capsule Frequency: Once a Day Duration: 60 Days Mode of Usage: Take the capsule once a day with food
  Arms: Botanical Extract Standardised for Iron

SUMMARY:
A randomized, double-blind, parallel, three-arms, placebo-controlled, safety and efficacy study of Botanical Extract Standardized for Iron + Vitamin C and Botanical Extract Standardized for Iron in adult human subjects with anemia or iron-deficiency anemia.

A total of up to 96 adult male and female subjects of age 26 to 55 years (32 subjects/arm) will be enrolled to get 90 evaluable subjects (30 subjects/arm) in the study

DETAILED DESCRIPTION:
The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The adult female/male subjects will be instructed to visit the facility as per the below visits. There will be total of 4 visits in this study.

* Visit 01 (Within 30 Days): Screening procedure, informed consent obtain process, baseline evaluations, blood collection, urine collection.
* Visit 02 (Day 01): Enrolment, randomization, product distribution, subject diary distribution, blood collection.
* Visit 03 (Day 30 ± 2 Days): Treatment period, blood collection, evaluations, consumer's QoL product perception questionnaire, subject diary review, AE reporting (if any).
* Visit 04 (Day 60 ± 2 Days): End of study process, evaluation, blood collection, urine collection, consumer's QoL and product perception questionnaire, subject diary collection, test treatments accountability, AE reporting (if any).

Assessment of efficacy parameters before test treatment usage will be done on screening visit within 30 days of Day 01, on Day 01 and after test treatment usage will be done on Day 30 (± 2 Days) and Day 60 (± 2 Days).

Blood Parameter Analysis: Hemoglobin, Hematocrit, RBC, WBC, MCV, MCH, MCHC, Serum Iron, Serum ferritin, Transferrin, Transferrin Saturation, Total Iron Binding Capacity, Total Cholesterol, Triglycerides, Random Glucose, Serum Creatinine, Uric Acid, SGPT, SGOT, LDL, HDL, HBsAG, SOD.

Urine Parameter: Chemical Parameters - Albumin, Blood, Glucose, pH; Physcial Parameters - Colour, Appearance and Deposits.

QoL Product Perception: Fatigue, Mood, Sleepiness, GI Discomfort, Energy Level, Epigastric Discomfort, Nausea, Diarrhoea, Constipation

ELIGIBILITY:
Inclusion Criteria:

1. Age: 26 to 55 years (both inclusive) at the time of consent.
2. Sex: Healthy males and non-pregnant/non-lactating females.
3. Subject suffering from iron deficiency anaemia of mild to moderate type (Hb range of 8-11mg/dl)
4. Subject must have negative Hepatitis B Surface Antigen (HBsAG)Test at screening.
5. Females of childbearing potential must have a reported negative urine pregnancy test.
6. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
7. Subject able to remain on stable usages of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
8. Subject able to forgo changes in baseline medications and nutritional supplements during the study period.
9. Subjects are willing to give written informed consent and are willing to follow the study procedure.
10. Subjects who commit not to use prescribed or OTC medication containing iron supplements for treatment of iron deficiency or anemia except test treatments for the entire duration of the study.
11. Subjects who are willing to use test treatments throughout the study period.

Exclusion Criteria:

1. Subject having other blood disease or any malignancy.
2. Subject with severe anemia (Hb < 8mg/dl).
3. Subject having any other chronic illness.
4. Subject with history of allergy or sensitivity to the test treatment ingredients.
5. Subject has a history of alcohol or drug addiction.
6. Any other condition which could warrant exclusion from the study, as per the investigator's discretion.
7. Pregnant or breastfeeding or planning to become pregnant during the study period.
8. Subject with history of acute blood loss.
9. Subject having a history of surgery in last 3-6 months.
10. Subjects participating in other similar nutraceuticals, food, supplemental or therapeutic trials within the last four weeks.

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Change in Haemoglobin [unit g/dl] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in haemoglobin in blood sample
Change in Haematocrit [unit %] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in haematocrit in blood sample
Change in RBC [unite 10^6/μl] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in RBC in blood sample
Change in serum iron [unite μg/dL] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in serum iron in blood sample
Change in serum ferritin level [unite μg/L] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in serum ferritin level in blood sample

SECONDARY OUTCOMES:
Change in transferrin [unite mg/dL] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in transferrin in blood sample
Change in transferrin saturation [unite %] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in transferrin saturation in blood sample
Change in iron binding capacity level [unite μg/dL] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in iron binding capacity in blood sample
Change in WBC count [unite 10^9/μl] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in WBC count in blood sample
Change in SOD level [unite U/ml] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change SOD level in blood sample
QOL product perception questionnaire | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of treatment perception by using 9-point hedonic scale
Change in CBC value [unite 10^6/μL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change CBC value in blood sample
Abnormal change in iron status | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of abnormal change iron status in blood sample
Change in total serum cholesterol [unite mg/dL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in total serum cholesterol level in blood sample
Change in triglyceride [unite mg/dL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in triglycerides in blood sample
Change in random blood glucose [unite mg/dL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in random blood glucose in blood sample
Change in serum creatinine [unite mg/dL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in serum creatinine in blood sample
Change in uric acid [unite mg/dL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in uric acid in blood sample
Change in SGPT [unite U/L] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in SGPT in blood sample
Change in SGOT [unite U/L] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in SGOT in blood sample
Change in LDL level [unite mg/dL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in LDL in blood sample
Change in HDL [unite mg/dL] | From baseline on screening visit before Day 01, before usage of test treatments on Day 01 and post-usage of test treatments on Day 30 (± 2 Days) and Day 60 (± 2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in HDL in blood sample
Abnormal change in presence of albumin [unite g/dL] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of abnormal change in presence of albumin in urine sample
Change in blood glucose [unite mg/dL] | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in blood glucose in urine sample
Change in urine pH | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in urine pH in urine sample
Change in colour of urine | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in colour of urine
Change in appearance of urine | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in appearance of urine
Change in deposits | From Baseline on Day 01 before usage of test treatments and post-usage of test treatments on Day 30 (+2 Days) and Day 60 (+2 Days) and compare with placebo arm
  To assess the effectiveness of the test treatment in terms of change in deposits in urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, Principal Investigator — Medical Direcor
Locations (1):
- NovoBliss Research Pvt.Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No